CLINICAL TRIAL: NCT02495428
Title: Effect of Kinesio Taping in Muscle Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEU-010
Record Dates: First submitted 2015-07-03; First posted 2015-07-13 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Muscle Fatigue
Keywords: Bandage; Treadmill; Lactate Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kinesio Tape Group (Experimental): muscle Kinesio Taping in Triceps Surae, Tibialis anterior, and Quadriceps according Kenzo Kase Method
  Interventions: Procedure: Kinesio Tape Method
- Control group (No Intervention): They will do the same measurement of lactate and exercise protocol in treadmill, but always without kinesio tape intervention

INTERVENTIONS:
Procedure: Kinesio Tape Method
  Arms: Kinesio Tape Group

SUMMARY:
The aim of this study was to determine the effect of Kinesio taping on lactic acid in an running anaerobic test.

ELIGIBILITY:
Inclusion Criteria:

* They should practice physical activity 2-4 days a week.

Exclusion Criteria:

* History of surgery in the lower limbs
* Muscle-tendon injury or trauma in the lower limbs (LL) in the last six months
* cardiovascular and / or respiratorydisease
* Any allergies related to the bandage material.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in capillary blood acid lactate | Participants will be measured four times to follow the changes of lactate: Baseline (Pre Exercise), immediately post exercise, 5 minutes post exercise and 15 minutes post exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- San Pablo CEU University, Boadilla del Monte, Madrid, Spain